CLINICAL TRIAL: NCT01756456
Title: An 8-week Phase I/II, Multicenter, Randomized, Double-masked, Vehicle Controlled Parallel Group Study to Evaluate the Safety and Efficacy of Two Doses of Recombinant Human Nerve Growth Factor in Patients With Stage 2 and 3 of NK
Brief Title: Evaluation of Safety and Efficacy of rhNGF in Patients With Stage 2 and 3 Neurotrophic Keratitis.
Acronym: REPARO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF0212; 2012-002527-15 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2017-02

CONDITIONS: Neurotrophic Keratitis; Keratitis; Corneal Ulcer
Keywords: Keratitis; Corneal Ulcer
MeSH Terms: conditions — Keratitis; Corneal Ulcer | interventions — cenegermin; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1_rhNGF10_Phase 1_treatment (Experimental): active treatment with rhNGF 10 μg/ml. One drop six times a day (one 35 μl drop equals to 0.35μg of rhNGF).
  Interventions: Drug: rhNGF 10 μg/ml
- 2_rhNGF20_Phase 1_treatment (Experimental): active treatment with rhNGF 20 μg/ml. One drop 6 times a day (one 35 μl drop equals to 0.70 μg of rhNGF)
  Interventions: Drug: rhNGF 20 μg/ml
- 3_vehicle group_Phase 1_treatment (Placebo Comparator): vehicle control arm. Ophthalmic solution of the same composition as the test product with the exception of rhNGF. One drop six times a day for the entire period
  Interventions: Other: vehicle
- 4_rhNGF10_Phase 2_treatment (Experimental): active treatment with rhNGF 10 μg/ml. One drop six times a day (one 35 μl drop equals to 0.35 μg of rhNGF)
  Interventions: Drug: rhNGF 10 μg/ml
- 5_rhNGF20_Phase 2_treatment (Experimental): active treatment with rhNGF 20 μg/ml. One drop 6 times a day (one 35 μl drop equals to 0.70 μg of rhNGF)
  Interventions: Drug: rhNGF 20 μg/ml
- 6_vehicle group_Phase 2_treatment (Placebo Comparator): vehicle control arm. Ophthalmic solution of the same composition as the test product with the exception of rhNGF. One drop six times a day for the entire period
  Interventions: Other: vehicle

INTERVENTIONS:
Drug: rhNGF 10 μg/ml — rhNGF 10 μg/ml : one drop 6 times a day (one 35 μl drop equals to 0.35 μg of rhNGF)
  Other Names: recombinant human nerve growth factor 10 µg/ml solution
  Arms: 1_rhNGF10_Phase 1_treatment; 4_rhNGF10_Phase 2_treatment
Drug: rhNGF 20 μg/ml — one drop 6 times a day (one 35 μl drop equals to 0.70 μg of rhNGF)
  Other Names: recombinant human nerve growth factor 20 µg/ml solution
  Arms: 2_rhNGF20_Phase 1_treatment; 5_rhNGF20_Phase 2_treatment
Other: vehicle — ophthalmic solution of the same composition as the test product without rhNGF
  Other Names: placebo
  Arms: 3_vehicle group_Phase 1_treatment; 6_vehicle group_Phase 2_treatment

SUMMARY:
This study is aimed at assessing the safety and the efficacy of two dose regimens of recombinant human nerve growth factor (rhNGF) eye drops solution compared to vehicle for inducing a complete healing of stage 2 (persistent epithelial defect) and 3 (corneal ulcer) neurotrophic keratitis

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and the efficacy of two dose regimens (10 µg/ml or 20 µg/ml 6 times a day) of recombinant human nerve growth factor (rhNGF) eye drops solution compared to vehicle for inducing a complete healing of stage 2 (persistent epithelial defect) and 3 (corneal ulcer) neurotrophic keratitis (NK) as measured by the Reading Center evaluating the clinical pictures of corneal fluorescein staining.

Secondary objectives of the study are to assess the duration of complete healing, improvement in visual acuity and improvement in corneal sensitivity following treatment with rhNGF eye drops solution

This is a combined phase I/II study. The phase I and II segments of the study will be conducted as an 8 week, randomized, double-masked, vehicle controlled, parallel group study (referred to as the controlled treatment period) followed by a 48 or 56 week follow-up period The design of the phase I and phase II segments of the study are identical with the exception that in the phase I segment of the study the randomization scheme is different and patients will be followed with additional safety assessments and blood samples for PK (pharmacokinetic) profiling In the ascending dose Phase I segment of the study two doses of rhNGF 10 and 20 µg/ml will be evaluated in a sequential manner

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Patients with stage 2 (persistent epithelial defect, PED) or stage 3 (corneal ulcer) neurotrophic keratitis involving only one eye. . Patients with Controlateral eye affected with stage 1 NK can be enrolled.
3. PED or corneal ulceration of at least 2 weeks duration refractory to one or more conventional non-surgical treatments for neurotrophic keratitis (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops and medications that can decrease corneal sensitivity; therapeutic contact lenses).
4. Evidence of decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet aesthesiometer) within the area of the PED or corneal ulcer and outside of the area of the defect in at least one corneal quadrant.
5. Best corrected distance visual acuity (BCDVA) score ≤ 75 ETDRS letters, (≥ 0.2 LogMAR, ≤ 20/32 Snellen or ≤ 0.625 decimal fraction) in the affected eye.
6. No objective clinical evidence of improvement in the PED or corneal ulceration within the 2 weeks prior to study enrolment.
7. Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representative must have been approved by the IEC/IRB for the current study.
8. Patients must have the ability and willingness to comply with study procedures.
9. Patients must be eligible for the National Health Insurance (where applicable).

Exclusion Criteria:

1. Patients with stage 2 or 3 NK affecting both eyes.
2. Any active ocular infection (bacterial, viral, fungal or protozoal) or active ocular inflammation not related to NK in the affected eye.
3. Any other ocular disease requiring topical ocular treatment in the affected eye during the course of the study treatment period. No topical treatments other than the study medications provided by the study sponsor or allowed by the study protocol can be administered in the affected eye during the course of the study treatment periods.
4. Patients with severe vision loss in the affected eye with no potential for visual improvement in the opinion of the investigator as a result of the study treatment.
5. Schirmer test without anesthesia ≤3 mm/5 minutes in the affected eye.
6. Patients with severe blepharitis and/or severe meibomian gland disease in the affected eye.
7. History of any ocular surgery (including laser or refractive surgical procedures) in the affected eye within the three months before study enrolment. (An exception to the preceding statement will be allowed if the ocular surgery is considered to be the cause of the stage 2 or 3 NK). Ocular surgery in the affected eye will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period.
8. Prior surgical procedure(s) for the treatment of NK (e.g. complete tarsorraphy, conjunctival flap, etc) in the affected eye with the exception of amniotic membrane transplantation. Patients previously treated with amniotic membrane transplantation may only be enrolled two weeks after the membrane has disappeared within the area of the PED or corneal ulcer or at least six weeks after the date of the amniotic membrane transplantation procedure. Patients previously treated with Botox (botulinum toxin) injections used to induce pharmacologic blepharoptosis are eligible for enrolment only if the last injection was given at least 90 days prior to enrolment in the study.
9. Use of therapeutic contact lenses or contact lens wear for refractive correction during the study treatment periods in the eye with NK.
10. Anticipated need for punctual occlusion during the study treatment period. Patients with punctual occlusion or punctual plugs inserted prior to the study are eligible for enrolment provided that the punctual occlusion is maintained during the study.
11. Evidence of corneal ulceration involving the posterior third of the corneal stroma, corneal melting or perforation in the affected eye.
12. Presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct (e.g. progressive or degenerative corneal or retinal conditions, uveitis, optic neuritis, poorly controlled diabetes, autoimmune disease, systemic infection, neoplastic diseases).
13. Any need for or anticipated change in the dose of systemic medications known to impair the function of the trigeminal nerve (e.g. neuroleptics, antipsychotic and antihistamine drugs). These treatments are allowed during the study if initiated prior to 30 days before study enrolment provided they remain stable throughout the course of the study treatment periods.
14. Known hypersensitivity to one of the components of the study or procedural medications (e.g. fluorescein).
15. History of drug, medication or alcohol abuse or addiction.
16. Use of any investigational agent within 4 weeks of screening visit.
17. Participation in another clinical study at the same time as the present study.
18. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions: are currently pregnant or have a positive result on the urine pregnancy test at the Randomization Visit or intend to become pregnant during the study treatment period or are breast-feeding or not willing to use highly effective birth control measures, such as: Hormonal contraceptives -oral, implanted, transdermal, or injected and/or Mechanical barrier methods -spermicide in conjunction with a barrier such as a condom or diaphragm or IUD during the entire course of and 30 days after the study treatment periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sinigaglia, MD, Study Director — Dompé s.p.a., Milan
Locations (34):
- France (5):
  - CHU de Dijon - Service ophtalmologie, Dijon
  - CHU Dupuytren - Service Ophtalmologie, Limoges
  - Centre Hospitalier National d'Ophtalmologie - Service d'ophtalmologie, Paris
  - "Fondation Ophtalmologique Adolphe de Rothschild - "Unité de Recherche Clinique, Paris
  - "CHU Toulouse-Purpan - Service Ophtalmologie, Toulouse
- Germany (6):
  - Universität zu Köln - Zentrum für Augenheilkunde am Universitätsklinikum Köln, Cologne
  - University Eye Clinic in Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitäts-Augenklinik Freiburg, Freiburg im Breisgau
  - Johannes-Gutenberg-Universität Augenklinik und Poliklinik - Department of Ophthalmology, Mainz
  - Klinikum der Universität München - Augenklinik der Ludwig-Maximilians-Universtiät München, München
- Italy (9):
  - OSPEDALE SAN RAFFAELE di Milano, Milan, Lombardy
  - Università G. D' Annunzio - Clinica Oftalmologica - Centro regionale di Eccellenza in Oftalmologia, Chieti
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Dipartimento di Scienze Neurologiche Oftalmologia e Genetica - Universtità di Genova, Genoa
  - Azienda Ospedaliero Universitaria di Messina - Dipartimento Specialità Chirurgiche Ambulatorio Studio delle Malattie dela Superficie Oculare Unità Operativa Complessa di Oftalmologia, Messina
  - Azienda Ospedaliera San Paolo - U.O. Oculistica, Milan
  - Azienda ospedaliera di Padova - Clinica Oculistica Policlinico 7° Piano, Padua
  - Università Campus Bio-Medico di Roma, Rome
  - Policlinico Umberto I, Rome
- Poland (2):
  - District Railway Hospital Katowice - Department of Ophthalmology, Katowice
  - "SPKSO Szpital Okulistyczny ul. - SPKSO Szpital Okulistyczny, Warsaw
- Spain (7):
  - Vissum Corporación Oftalmológica de Alicante, Alicante
  - Hospital de Cruces - Oftalmología, Barakaldo
  - Barraquer Eye center, Barcelona
  - Hospital Clinic de Barcelona - Oftalmología, Barcelona
  - Hospital Clínico San Carlos - Oftalmología. Unidad de Superficie Ocular, Madrid
  - Instituto Oftalmológico Fernández-Vega - Oftalmología, Oviedo
  - Cartuja Visión - Oftalmología, Seville
- United Kingdom (5):
  - University of Birmingham - Academic Unit of Ophthalmology, School of Immunity and Infection, College of Medical and Dental Sciences, University of Birmingham, Birmingham
  - Moorfields Eye Hospital - Moorfields Eye Hospital, London
  - Manchester Royal Eye Hospital - Manchester Royal Eye Hospital, Manchester
  - Royal Victoria Infirmary - Dept. of Ophthalmology, Newcastle upon Tyne
  - University of Southampton Southampton General Hospital - MP104, Eye Unit, Southampton

REFERENCES:
- [Derived] Yanai R, Nishida T, Chikama T, Morishige N, Yamada N, Sonoda KH. Potential New Modes of Treatment of Neurotrophic Keratopathy. Cornea. 2015 Nov;34 Suppl 11:S121-7. doi: 10.1097/ICO.0000000000000587. PMID 26448169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 periods: 8week PhaseI/controlled treatment period and 48/56-week FU period. In the Phase1 patients were randomized into 2 cohorts (of 9 pts each). In phase 2 pts were randomized in a 1:1:1 ratio (52 pts each group). Data refer to the 1st database lock when the last patient in Phase2 had completed 12 weeks of FU period.
Pre-assignment Details: The inclusion/exclusion criteria were designed to include individuals 18 years of age or older with Stage 2 (PED) or Stage 3 (corneal ulcer) NK involving only 1 eye and to exclude those with Stage 2 or 3 NK affecting both eyes, any active ocular infection or inflammation not related to NK, or any ocular disease or severe vision loss.
Groups:
- 1_rhNGF 10µg/ml Phase 1_treatment: rhNGF 10 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 2_rhNGF 20 µg/ml_Phase 1_treatment: rhNGF 20 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 3_vehicle group_Phase 1_treatment: Placebo eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
Period: Treatment Period: Phase I/II
Arm/Group | 1_rhNGF 10µg/ml Phase 1_treatment | 2_rhNGF 20 µg/ml_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Started | 7 | 7 | 4 | 52 | 52 | 52
Completed | 6 | 6 | 2 | 45 | 39 | 48
Not Completed | 1 | 1 | 2 | 7 | 13 | 4
Not completed — decision unrelated to adverse event | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 3 | 9 | 1
Not completed — Other causes | 0 | 0 | 0 | 1 | 2 | 2
Period: Follow Up Period Phase I/II
Arm/Group | 1_rhNGF 10µg/ml Phase 1_treatment | 2_rhNGF 20 µg/ml_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Started | 6 | 6 | 2 | 45 | 39 | 48
Completed | 5 | 5 | 1 | 12 | 13 | 15
Not Completed | 1 | 1 | 1 | 33 | 26 | 33
Not completed — still in study after week 20 | 0 | 0 | 0 | 25 | 23 | 25
Not completed — parent withdrew the consent to continue | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 5 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Other causes | 0 | 0 | 0 | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- 1_rhNGF10_Phase 1_treatment: rhNGF 10 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 2_rhNGF20_Phase 1_treatment: rhNGF 20 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 4_rhNGF10_Phase 2_treatment: rhNGF 10 µg/ml eye drops solution: rhNGF 10 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 5_rhNGF20_Phase 2_treatment: rhNGF 20 µg/ml eye drops solution: rhNGF 20 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 6_vehicle group_Phase 2_treatment: Placebo: Placebo eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only.
- Total: Total of all reporting groups
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment | Total
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The patients populations of Phase I and Phase II are different. The first consists of 18 individuals, the second of 156 individuals.
  years
    Age continuous | 61.7 (21.47) | 52.0 (17.24) | 64.3 (24.06) | 59.0 (17.17) | 62.5 (14.01) | 60.4 (16.78) | 58.5 (19.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 30 | 30 | 35 | 104
  Male | 4 | 3 | 2 | 22 | 22 | 17 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 6 | 9 | 5 | 21
  Not Hispanic or Latino | 6 | 6 | 4 | 42 | 42 | 41 | 141
  Unknown or Not Reported | 0 | 1 | 0 | 4 | 1 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Healing of the Persistent Epithelial Defect (PED) or Corneal Ulcer
Description: Complete healing of the PED or corneal ulcer was determined by corneal fluorescein staining at 4 weeks as defined by the reading center evaluating the clinical pictures.
  Complete healing was defined as the greatest diameter of the corneal fluorescein staining in the area of the PED or corneal ulcer being less than 0.5 mm at the Week 4 visit.
  The primary efficacy variable was analyzed after 4 weeks of treatment only for the Phase II segment of the study. That's why the Phase I groups/arms are not included in this analysis.
Time Frame: at 4 weeks of treatment
Population: Phase II patients who achieved complete healing at Week 4 (last observation carried forward - LOCF) as determined by the reading center (ITT population).
Measure: Number; unit: percentage of subjects
Arm/Group | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 52 | 52 | 52
percentage of subjects
  Yes | 55 | 58 | 20
  No | 45 | 42 | 80
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Phase II; Test type: Superiority — Each of the comparisons was conducted on the data for the Phase II segment of the study using a 2 × 2 chi-square test, based on the null hypothesis that there is no association between treatment (rhNGF or Vehicle Control) and response (Complete Healing at Week 4 [Yes/No]); p < 0.001, Chi-squared; Difference in percentage = 35.3, 97.06% CI 2-sided [15.88 to 54.71]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, Chi-squared; Difference in percentage = 38.4, 97.06% CI 2-sided [18.96 to 57.83]

2. Secondary Outcome: Percentage of Patients Experiencing Healing of the Persistent Epithelial Defect (PED) or Corneal Ulcer
Description: Complete healing of the PED or corneal ulcer at 4 weeks as defined by the Investigator. The complete healing was defined as the greatest diameter of the corneal fluorescein staining in the area of the PED or corneal ulcer, being less than 0.5 mm at the Week 4 visit.
  This secondary outcome was analyzed after 4 weeks of treatment only for the Phase II segment of the study. That's why the Phase I groups/arms are not included in this analysis.
Time Frame: at 4 weeks of study treatment.
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 52 | 52 | 52
percentage of subjects
  Yes | 52 | 61 | 26
  No | 48 | 39 | 74
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority; p = 0.016, Chi-squared; Difference in percentage = 25.8, 97.06% CI 2-sided [3.66 to 47.87]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority; p = 0.002, Chi-squared; Difference in percentage = 34.7, 97.06% CI 2-sided [11.91 to 57.41]

3. Secondary Outcome: Percentage of Patients Experiencing Complete Healing of the Persistent Epithelial Defect (PED) or Corneal Ulcer
Description: Complete healing of the PED or corneal ulcer at 6 and 8 weeks measured by both the central reading center and Investigator.
  Complete healing was defined as the greatest diameter of the corneal fluorescein staining in the area of the PED or corneal ulcer being less than 0.5 mm.
  This outcome was analyzed after 6 and 8 weeks of treatment only for the Phase II segment of the study. That's why the Phase I groups/arms are not included in this analysis.
Time Frame: at 6 and 8 weeks after start of the treatment
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 52 | 52 | 52
percentage of subjects
  week 6 - central reading center - yes | 68 | 60 | 66
  week 6 - central reading center - no | 32 | 40 | 34
  week 6 - investigator - yes | 61 | 64 | 41
  week 6 - investigator - no | 39 | 36 | 59
  week 8 - central reading center - yes | 78 | 83 | 56
  week 8 - central reading center - no | 22 | 17 | 44
  week 8 - investigator - yes | 79 | 79 | 53
  week 8 - investigator - no | 21 | 21 | 47
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; At week 6 - reading center; Test type: Superiority; p = 0.818, Chi-squared; difference in percentage = 2.4, 97.06% CI 2-sided [-20.30 to 25.08]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; at week 6 - central reading center; Test type: Superiority; p = 0.571, Chi-squared; difference in percentage = -6.3, 97.06% CI 2-sided [-30.62 to 17.96]
Statistical Analysis 3: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6 - investigator; Test type: Superiority; p = 0.064, Chi-squared; Difference in percentage = 20.3, 97.06% CI 2-sided [-3.11 to 43.79]
Statistical Analysis 4: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6 - investigator; Test type: Superiority; p = 0.041, Chi-squared; Difference in percentage = 23.1, 97.06% CI 2-sided [-0.89 to 47.04]
Statistical Analysis 5: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8 - central reading center; Test type: Superiority; p = 0.031, Chi-squared; Difference in percentage = 21.9, 97.06% CI 2-sided [0.07 to 43.64]
Statistical Analysis 6: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8 - central reading center; Test type: Superiority; p = 0.008, Chi-squared; difference in percentage = 26.9, 97.06% CI 2-sided [5.57 to 48.28]
Statistical Analysis 7: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8 - investigator; Test type: Superiority; p = 0.011, Chi-squared; Difference in percentage = 26.1, 97.06% CI 2-sided [4.18 to 48.01]
Statistical Analysis 8: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8 - investigator; Test type: Superiority; p = 0.014, Chi-squared; Difference in percentage = 25.9, 97.06% CI 2-sided [3.55 to 48.33]

4. Secondary Outcome: Percentage of Patients Experiencing Complete Corneal Clearing
Description: Complete corneal clearing (grade 0 on the modified Oxford scale) at 4, 6 and 8 weeks.
  A patient was considered to have achieved complete corneal clearing if he/she had a Modified Oxford Scale recorded as Grade 0.
  The scale has the following grades: 0-1-2-3-4-5, where 5 represents the worst outcome value and 0 the best outcome value.
Time Frame: at 4, 6 and 8 weeks after start of the treatment
Population: ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of subjects
  week 4 - yes | 0 | 17 | 33 | 21 | 20 | 7
  week 4 - no | 100 | 83 | 67 | 79 | 80 | 93
  week 6 - yes | 17 | 14 | 0 | 24 | 23 | 8
  week 6 - no | 83 | 86 | 100 | 76 | 77 | 92
  week 8 -yes | 17 | 14 | 0 | 27 | 21 | 10
  week 8 - no | 83 | 86 | 100 | 73 | 79 | 90
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.065, Chi-squared; difference in percentage = 13.7, 95% CI 2-sided [-0.19 to 27.57]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.097, Chi-squared; difference in percentage = 12.4, 95% CI 2-sided [-2.05 to 26.78]
Statistical Analysis 3: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.036, Chi-squared; difference in percentage = 16.9, 95% CI 2-sided [1.97 to 31.92]
Statistical Analysis 4: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.054, Chi-squared; difference in percentage = 15.6, 95% CI 2-sided [0.04 to 31.12]
Statistical Analysis 5: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.043, Chi-squared; difference in percentage = 17.1, 95% CI 2-sided [1.45 to 32.72]
Statistical Analysis 6: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.157, Chi-squared; difference in percentage = 11.4, 95% CI 2-sided [-4.08 to 26.93]

5. Secondary Outcome: Mean Change in Best Corrected Distance Visual Acuity (BCDVA)
Description: Mean changes in Best-Corrected Distance Visual Acuity (BCDVA) from baseline to Week 8 are calculated as Least Square means. BCDVA consists of letters read at 4 meters only. Patients are scored by how many letters could be correctly identified. Therefore the higher the number of letters, the higher the visual acuity.
Time Frame: At screening and at week 8
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: LogMAR
Arm/Group | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 52 | 52 | 52
LogMAR | 15.8 (2.58) | 11.9 (2.80) | 6.9 (2.83)
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority; p = 0.022, ANCOVA; least square mean difference = 8.9, 95% CI 2-sided [1.33 to 16.50]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority; p = 0.213, ANCOVA; least square mean difference = 5.0, 95% CI 2-sided [-2.90 to 12.88]

6. Secondary Outcome: Percentage of Patients That Achieve an Improvement in Corneal Sensitivity
Description: Percentage of patients that achieve an improvement in corneal sensitivity as measured by the Cochet-Bonnet aesthesiometer
Time Frame: at 4, 6 and 8 weeks.
Population: ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of subjects
  week 4 - yes | 67 | 50 | 50 | 69 | 61 | 63
  week 4 - no | 33 | 50 | 50 | 31 | 39 | 37
  week 6 - yes | 67 | 50 | 50 | 83 | 68 | 55
  week 6 - no | 33 | 50 | 50 | 17 | 32 | 45
  week 8 -yes | 67 | 60 | 100 | 79 | 76 | 68
  week 8 - no | 33 | 40 | 0 | 21 | 24 | 32
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.592, Chi-squared; difference in percentage = 5.5, 95% CI 2-sided [-14.53 to 25.48]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority — week 4; p = 0.835, Chi-squared; difference in percentage = -2.3, 95% CI 2-sided [-24.01 to 19.40]
Statistical Analysis 3: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.008, Chi-squared; difference in percentage = 27.7, 95% CI 2-sided [8.10 to 47.22]
Statistical Analysis 4: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.282, Chi-squared; difference in percentage = 12.4, 95% CI 2-sided [-9.91 to 34.68]
Statistical Analysis 5: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; Test type: Superiority; p = 0.303, Chi-squared; difference in percentage = 10.2, 95% CI 2-sided [-9.15 to 29.45]
Statistical Analysis 6: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.442, Chi-squared; difference in percentage = 7.9, 95% CI 2-sided [-12.13 to 27.92]

7. Secondary Outcome: Percentage of Patients Experiencing Deterioration in Stage 2 or 3 NK
Description: Percentage of patients experiencing deterioration (increase in lesion size ≥ 1mm, decrease in BCDVA by >5 ETDRS letters, progression in lesion depth to corneal melting or perforation, onset of infection) in stage 2 or 3 NK from baseline to Week 4, 6, and 8.
Time Frame: from baseline to Week 4, 6, and 8.
Population: ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of subjects
  week 4 - yes | 0 | 0 | 0 | 2 | 2 | 5
  week 4 - no | 100 | 100 | 100 | 98 | 98 | 95
  week 6 - yes | 0 | 0 | 0 | 2 | 0 | 10
  week 6 - no | 100 | 100 | 100 | 98 | 100 | 90
  week 8 -yes | 0 | 14 | 0 | 4 | 7 | 15
  week 8 - no | 100 | 86 | 100 | 96 | 93 | 85
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.597, Chi-squared; difference in percentage = -2.6, 95% CI 2-sided [-22.87 to 17.71]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p > 0.999, Chi-squared; difference in percentage = -2.3, 95% CI 2-sided [-23.26 to 18.71]
Statistical Analysis 3: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.183, Chi-squared; difference in percentage = -7.8, 95% CI 2-sided [-28.70 to 13.76]
Statistical Analysis 4: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.116, Chi-squared; difference in percentage = -10.0, 95% CI 2-sided [-31.41 to 11.88]
Statistical Analysis 5: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.134, Chi-squared; difference in percentage = -10.8, 95% CI 2-sided [-31.30 to 10.35]
Statistical Analysis 6: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.307, Chi-squared; difference in percentage = -7.9, 95% CI 2-sided [-29.51 to 13.52]

8. Secondary Outcome: Percentage of Patients Achieving Complete Healing of the PED or Corneal Ulcer by Week 8/16 That Remain Healed at Weeks 20/28, 32/40, 44/52, 56/64
Description: Percentage of patients achieving complete healing of the PED or corneal ulcer by Week 8/16 that remain healed (ie, no recurrence of the PED and/or corneal ulcer) at Weeks 20/28, 32/40, 44/52, 56/64
Time Frame: at week 20/28, 32/40, 44/52, and 56/64
Population: ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of subjects
  week 20/28 - yes | 100 | 75 | 100 | 87 | 89 | 100
  week 20/28 - no | 0 | 25 | 0 | 13 | 11 | 0
  week 32/40 - yes | 100 | 75 | 100 | 78 | 92 | 100
  week 32/40 - no | 0 | 25 | 0 | 22 | 8 | 0
  week 44/52 - yes | 100 | 80 | 100 | 67 | 88 | 100
  week 44/52 - no | 0 | 20 | 0 | 33 | 12 | 0
  week 56/64 - yes | 100 | 80 | 100 | 67 | 82 | 100
  week 56/64 - no | 0 | 20 | 0 | 33 | 18 | 0

9. Secondary Outcome: Percentage of Patients Experiencing a Different Level of Efficacy at 4 and 8 Weeks
Description: Global evaluation of efficacy as assessed by the Investigator at 4 and 8 weeks. The different level of efficacy were: very good; good; moderate; poor; non-evaluable.
Time Frame: at week 4 and 8
Population: ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of subjects
  week 4 - very good | 17 | 29 | 67 | 40 | 34 | 26
  week 4 - good | 33 | 43 | 0 | 38 | 49 | 35
  week 4 - moderate | 17 | 0 | 0 | 15 | 7 | 21
  week 4 - poor | 33 | 29 | 0 | 6 | 10 | 19
  week 4 - non-evaluable | 0 | 0 | 33 | 2 | 0 | 0
  week 8 - very good | 17 | 29 | 50 | 48 | 40 | 40
  week 8 - good | 33 | 43 | 50 | 31 | 45 | 20
  week 8 - moderate | 33 | 0 | 0 | 12 | 5 | 12
  week 8 - poor | 17 | 29 | 0 | 4 | 10 | 28
  week 8 - non-evaluable | 0 | 0 | 0 | 4 | 0 | 0
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.041, Chi-squared; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.03 to 4.62]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.081, Chi-squared; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.92 to 4.11]
Statistical Analysis 3: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.040, Chi-squared; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.04 to 5.88]
Statistical Analysis 4: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.132, Chi-squared; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.82 to 4.52]

10. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Ocular Tolerability
Description: Ocular tolerability was recorded by the patient on a VAS scale from 0 to 100 mm, where a higher VAS score indicates worse ocular symptoms (0 means no symptoms and 100 means the worst possible discomfort). The overall VAS score for ocular tolerability was calculated as the mean of the individual VAS scores for the 7 different symptoms (foreign body sensation, burning/stinging, itching, ocular pain, sticky feeling, blurred vision and photophobia).
  Results are below reported as per symptoms at week 8 (for treatment period) and week 20 (for Follow Up period).
Time Frame: at baseline and at weeks 8 and 20
Population: Safety population
Measure: Mean (Standard Deviation); unit: VAS score
Groups:
- 1_rhNGF10_Phase 1_FU: Follow up for Phase 1 active treatment with rhNGF 10 μg/ml
- 2_rhNGF20_Phase 1_FU: Follow up for Phase 1 active treatment with rhNGF 20 μg/ml
- 3_vehicle group_Phase 1_FU: Follow up for Phase 1 vehicle control arm
- 4_rhNGF10_Phase 2_FU: Follow up for Phase 2 active treatment with rhNGF 10 μg/ml
- 5_rhNGF20_Phase 2_FU: Follow up for Phase 2 active treatment with rhNGF 20 μg/ml
- 6_vehicle_Phase 2_FU: Follow up for Phase 2 vehicle control arm
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment | 1_rhNGF10_Phase 1_FU | 2_rhNGF20_Phase 1_FU | 3_vehicle group_Phase 1_FU | 4_rhNGF10_Phase 2_FU | 5_rhNGF20_Phase 2_FU | 6_vehicle_Phase 2_FU
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52 | 6 | 6 | 2 | 45 | 39 | 48
VAS score
  Foreign Body Sensation_Baseline | 50.4 (25.68) | 24 (19.76) | 20.5 (29.23) | 34.8 (29.4) | 35.4 (34.79) | 37.7 (36.49) | 50.4 (25.68) | 24 (19.76) | 20.5 (29.23) | 34.8 (29.4) | 35.4 (34.79) | 37.7 (36.49)
  Foreign Body Sensation_CFB | -21.2 (25.96) | -12.9 (17.03) | -16 (65.05) | -8.8 (34.68) | -16.5 (36.87) | -20.9 (35.86) | -20 (30.32) | -13 (25.3) | -52 (0) | -16.6 (31.26) | -22.4 (38.77) | -20.7 (30.57)
  burning/stinging_baseline | 41.4 (30.85) | 30.7 (38.78) | 18 (28.57) | 32.5 (32.88) | 26.5 (30.86) | 30.2 (32.21) | 41.4 (30.85) | 30.7 (38.78) | 18 (28.57) | 32.5 (32.88) | 26.5 (30.86) | 30.2 (32.21)
  burning/stinging_CFB | -14.7 (38.02) | -12.1 (28.27) | -28.5 (23.33) | -3.8 (42.13) | -2.5 (26.76) | -18 (32.97) | -18 (41.65) | -16.5 (17.13) | -12 (0) | -14.9 (40.35) | -10.8 (31.51) | -14.7 (37.54)
  itching_baseline | 17 (27.4) | 18.7 (19.62) | 7.8 (15.5) | 24.1 (27.48) | 21.8 (28.68) | 22.9 (28.43) | 17 (27.4) | 18.7 (19.62) | 7.8 (15.5) | 24.1 (27.48) | 21.8 (28.68) | 22.9 (28.43)
  itching_CFB | -3 (17.93) | -10 (23.1) | -15.5 (21.92) | -10.8 (29.25) | -7.3 (22.67) | -8.9 (25.59) | -7.8 (27.18) | -4.2 (28.51) | -31 (0) | -10.2 (30.62) | -11.9 (23.05) | -4.8 (30.71)
  ocular pain_baseline | 34.1 (36.96) | 33.6 (34.73) | 19 (38) | 32.8 (34.86) | 21.1 (28.38) | 28.8 (32.82) | 34.1 (36.96) | 33.6 (34.73) | 19 (38) | 32.8 (34.86) | 21.1 (28.38) | 28.8 (32.82)
  ocular pain_CFB | -21.2 (28.96) | -6 (30.72) | -23 (32.53) | -2 (43) | 2 (37.25) | -16.3 (30.52) | -16 (28.59) | -9.3 (11.86) | -26 (0) | -16.7 (34.66) | -12.1 (31.25) | -18.3 (34.3)
  sticky feeling_baseline | 47.6 (34.14) | 32.1 (35.34) | 15.5 (23.69) | 26.6 (29.65) | 17.4 (22.07) | 26.1 (31.93) | 47.6 (34.14) | 32.1 (35.34) | 15.5 (23.69) | 26.6 (29.65) | 17.4 (22.07) | 26.1 (31.93)
  sticky feeling_CFB | -7.2 (42.82) | -18.7 (38.32) | -11 (5.66) | -11.7 (30.17) | -4.3 (29.55) | -10.7 (29.95) | -19.8 (22.18) | -0.7 (12.52) | -2 (0) | -13.3 (30.75) | -11.4 (31.11) | -8.3 (30.62)
  blurred vision_baseline | 71 (38.37) | 85.7 (14.74) | 93.5 (7.9) | 80.2 (25.18) | 83.2 (24.45) | 78.5 (24.68) | 71 (38.37) | 85.7 (14.74) | 93.5 (7.9) | 80.2 (25.18) | 83.2 (24.45) | 78.5 (24.68)
  blurred vision_CFB | -25.7 (34.37) | -25 (32.15) | -22 (31.11) | -24.9 (35.33) | -26.2 (31.58) | -17.4 (28.55) | -26.5 (31.18) | -26.2 (17.93) | -14 (0) | -16.5 (38.42) | -25.7 (34.41) | -17.4 (27.14)
  photophobia_baseline | 64.7 (42.9) | 66.6 (29.85) | 30.3 (26.21) | 64.3 (32.07) | 57.6 (36.1) | 65.2 (34.71) | 64.7 (42.9) | 66.6 (29.85) | 30.3 (26.21) | 64.3 (32.07) | 57.6 (36.1) | 65.2 (34.71)
  photophobia_CFB | -19.5 (27.98) | -20.7 (34.13) | -30.5 (43.13) | -17.8 (41.23) | -13.2 (40.44) | -17.5 (29.02) | -20.3 (28.63) | -26 (39.88) | -61 (0) | -24.2 (37.51) | -21 (38.76) | -14.6 (29.19)

11. Secondary Outcome: Change From Baseline in Best Corrected Distance Visual Acuity (BCDVA)
Description: Best-Corrected Distance Visual Acuity (BCDVA) by means of the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity chart at 4 meters (13 feet). Data reported refers to week n° 8 (treatment group) and n°12/20 (FU group).
Time Frame: at baseline and at period 1 (8 weeks) and 2 (Follow Up period of 12 weeks, until week 20)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Number of ETDRS letters
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment | 1_rhNGF10_Phase 1_FU | 2_rhNGF20_Phase 1_FU | 3_vehicle group_Phase 1_FU | 4_rhNGF10_Phase 2_FU | 5_rhNGF20_Phase 2_FU | 6_vehicle_Phase 2_FU
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52 | 6 | 6 | 2 | 45 | 39 | 48
Number of ETDRS letters
  Baseline | 42 (28.25) | 30.4 (24.85) | 9.5 (11.96) | 30.7 (28.35) | 24.2 (25.88) | 32.4 (26.07) | 42 (28.25) | 30.4 (24.85) | 9.5 (11.96) | 30.7 (28.35) | 24.2 (25.88) | 32.4 (26.07)
  Change from baseline | 9.3 (5.89) | 8.7 (12.41) | -1 (1.41) | 15.8 (16.82) | 11.9 (20.9) | 6.9 (15.44) | 11.2 (7.47) | 7 (9.8) | -6 (0) | 13.2 (16.8) | 14.2 (19.6) | 8.8 (14.27)

12. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP was measured using a Goldmann applanation tonometer, a handheld applanation tonometer [eg, Tonopen], or other tonometer, after the instillation of a topical anesthetic.
Time Frame: Baseline, period 1 (8 weeks) and 2 (Follow Up period of 12 weeks, until week 20).
Population: safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment | 1_rhNGF10_Phase 1_FU | 2_rhNGF20_Phase 1_FU | 3_vehicle group_Phase 1_FU | 4_rhNGF10_Phase 2_FU | 5_rhNGF20_Phase 2_FU | 6_vehicle_Phase 2_FU
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52 | 6 | 6 | 2 | 45 | 39 | 48
mmHg
  Baseline | 16.1 (3.85) | 11.3 (3.68) | 11.8 (3.3) | 14.3 (3.16) | 14 (3.06) | 14.1 (3.16) | 16.1 (3.85) | 11.3 (3.68) | 11.8 (3.3) | 14.3 (3.16) | 14 (3.06) | 14.1 (3.16)
  Change from baseline | -1.8 (2.48) | 1.9 (5.24) | 3.5 (2.12) | -0.1 (3.71) | 0.9 (2.61) | 0.8 (3.43) | -2.2 (2.49) | 2.3 (3.78) | -3 (0) | 0.2 (3.25) | 0.1 (3.64) | 0.6 (3.93)

13. Secondary Outcome: Percentage of Participants With Abnormal Eye Structures by Dilated Fundus Ophthalmoscopy
Description: Dilated fundus ophthalmoscopy was performed to assess the vitreous, retina, macula, choroid and optic nerve head after dilation of the pupil.
  Percentage of patients is summarized for each eye structure by treatment and visit for the controlled treatment period for Phase I and Phase II separately.
  The assessment time points were Baseline, weeks 2, 4 and 8 for Phase 1; Baseline and week 8 for Phase 2; and weeks 12 and 56 for follow up.
  Only results for eye structure at week 8 are reported.
Time Frame: At week 8 (Phase 1 and Phase 2)
Population: safety population
Measure: Number; unit: percentage of participants
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of participants
  Vitreous | 0 | 0 | 0 | 14.7 | 18.2 | 10.3
  Retina macula | 25 | 25 | 100 | 17.6 | 23.3 | 28.6
  Choroid | 0 | 25 | 0 | 8.8 | 6.5 | 14.8
  Optic nerve | 25 | 0 | 100 | 11.8 | 12.5 | 7.7

14. Other Pre Specified Outcome: Percentage of Patients That Achieved a ≥15 Letter Gain in BCDVA
Description: Percentage of patients that achieved a ≥15 letter gain in best corrected distance visual acuity (BCDVA) at 4, 6, and 8 weeks
Time Frame: at 4, 6 and 8 weeks
Population: ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | 1_rhNGF10_Phase 1_treatment | 2_rhNGF20_Phase 1_treatment | 3_vehicle group_Phase 1_treatment | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
Number analyzed (Participants) | 7 | 7 | 4 | 52 | 52 | 52
percentage of subjects
  week 4 - yes | 0 | 29 | 0 | 37 | 34 | 21
  week 4 - no | 100 | 71 | 100 | 63 | 66 | 79
  week 6 - yes | 17 | 43 | 0 | 44 | 38 | 28
  week 6 - no | 83 | 57 | 100 | 56 | 62 | 72
  week 8 -yes | 17 | 43 | 0 | 50 | 42 | 22
  week 8 - no | 83 | 57 | 100 | 50 | 58 | 78
Statistical Analysis 1: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.097, Chi-squared; difference in percentage = 15.8, 95% CI 2-sided [-2.36 to 33.97]
Statistical Analysis 2: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 4; Test type: Superiority; p = 0.175, Chi-squared; difference in percentage = 13.2, 95% CI 2-sided [-5.72 to 32.15]
Statistical Analysis 3: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.105, Chi-squared; difference in percentage = 16.9, 95% CI 2-sided [-3.11 to 37.00]
Statistical Analysis 4: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 6; Test type: Superiority; p = 0.300, Chi-squared; difference in percentage = 11.0, 95% CI 2-sided [-9.64 to 31.57]
Statistical Analysis 5: Comparison: 4_rhNGF10_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.008, Chi-squared; difference in percentage = 27.5, 95% CI 2-sided [8.33 to 46.67]
Statistical Analysis 6: Comparison: 5_rhNGF20_Phase 2_treatment vs 6_vehicle group_Phase 2_treatment; week 8; Test type: Superiority; p = 0.068, Chi-squared; difference in percentage = 19.0, 95% CI 2-sided [-0.91 to 38.83]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each time point of Phase I and Phase II of the study. Phase I: Days 1, 2, Weeks 1, 2, 3, 4, 6, Day 55, Week 8 Phase II: Weeks 1, 2, 3, 4, 6, 8
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information does not differ from the clinicaltrials.gov Definitions.
Groups:
- 1_rhNGF10_Phase 1: rhNGF 10 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 2_rhNGF20_Phase 1: rhNGF 20 µg/ml eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
- 3_vehicle group_Phase 1: Placebo eye drops solution, one drop 6 times a day for 8 weeks in the affected eye only
Arm/Group | 1_rhNGF10_Phase 1 | 2_rhNGF20_Phase 1 | 3_vehicle group_Phase 1 | 4_rhNGF10_Phase 2_treatment | 5_rhNGF20_Phase 2_treatment | 6_vehicle group_Phase 2_treatment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/4 | 5/52 | 2/52 | 1/52
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/7 | 3/4 | 13/52 | 14/52 | 4/52
Other Adverse Events (participants affected / at risk) | 3/7 | 5/7 | 1/4 | 23/52 | 23/52 | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1_rhNGF10_Phase 1 (N=7) | 2_rhNGF20_Phase 1 (N=7) | 3_vehicle group_Phase 1 (N=4) | 4_rhNGF10_Phase 2_treatment (N=52) | 5_rhNGF20_Phase 2_treatment (N=52) | 6_vehicle group_Phase 2_treatment (N=52)
disease progression (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Corneal graft rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal endotheliitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal epithelium defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurotrophic keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1_rhNGF10_Phase 1 (N=7) | 2_rhNGF20_Phase 1 (N=7) | 3_vehicle group_Phase 1 (N=4) | 4_rhNGF10_Phase 2_treatment (N=52) | 5_rhNGF20_Phase 2_treatment (N=52) | 6_vehicle group_Phase 2_treatment (N=52)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 | 2 (2) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Corneal graft rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 4 (6) | 6 (6)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Instillation site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vital dye staining cornea present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 3 (6) | 1 (2) | 2 (2) | 7 (7) | 5 (7)
Eye inflammation (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Corneal epithelium defect (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 1 (2)
Corneal lesion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Eyelid margin crusting (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Corneal decompensation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Ocular hyperemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 1 (2)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Lacrimation decreased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Corneal deposits (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Corneal endotheliitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lagophthalmos (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudopterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal cyst (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
Corneal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 1 (1)
Neurotrophic keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Conjunctivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis herpetic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blister infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Herpes simplex ophtalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster ophtalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No